CLINICAL TRIAL: NCT03027414
Title: The Effect of Transcranial Magnetic Stimulation to the Frontoparietal Attention Network on Anxiety Potentiated Startle
Brief Title: Effect of Transcranial Magnetic Stimulation to the Frontoparietal Attention Network on Anxiety Potentiated Startle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 170042; 17-M-0042
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
Keywords: Anxiety; Startle; Dorsolateral Prefrontal Cortex; Transcranial Magnetic Stimulation (TMS); Working Memory
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Substudy 1 Active and Sham (Experimental): HVs that receive TMS over the right dlPFC
  Interventions: Drug: Transcranial Magnetic Stimulation Sham; Device: Transcranial Magnetic Stimulation
- Substudy 2 Active and Sham (Experimental): HVs that receive TMS over the right dlFPC
  Interventions: Drug: Transcranial Magnetic Stimulation Sham; Device: Transcranial Magnetic Stimulation
- Substudy 3 Active and Sham (Experimental): HVs will receive offline TMS to the lest IPS (FPN)
  Interventions: Drug: Transcranial Magnetic Stimulation Sham; Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Drug: Transcranial Magnetic Stimulation Sham — TMS device is used to determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects.
Device: Transcranial Magnetic Stimulation — TMS device is used to determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects.

SUMMARY:
Background:

Researchers want to better understand brain processes related to fear and anxiety. They want to find out if transcranial magnetic stimulation (TMS), a type of brain stimulation, can reduce anxiety.

Objective:

To see how TMS affects fear and anxiety through memory and attention tasks.

Eligibility:

Healthy people ages 18-50 who are right-handed

Design:

Participants will be screened through another protocol.

Participants in the pilot study will have 1 visit. This includes:

Urine tests

Questionnaires about mood and thinking

Shock and startle workup: Electrodes are taped to the wrists or fingers. Participants will be shocked to find out what level of shock is uncomfortable but tolerable. They will hear loud, sudden noises through headphones.

TMS: A coil is held on the scalp. A magnetic field stimulates the brain. Sometimes they might receive fake TMS. This feels the same as real TMS. They will perform simple tasks. Participants in the main study will have 2 visits within 2 weeks.

The first visit includes:

Urine tests

Questionnaires about mood and thinking

MRI: Participants lie on a table that slides into a scanner. They will be in the scanner about 1 hour. A computer screen in the scanner will tell them to perform simple tasks.

The second visit includes:

Shock and startle workup

TMS

DETAILED DESCRIPTION:
Objective: To determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects. Toward this aim we will test the effect of transcranial magnetic stimulation (TMS) on two outcome measures: 1) Fear and anxiety during the threat of predictable and unpredictable shock (NPU threat test; Substudies 1 and 3), and 2) Working memory (WM) related anxiety downregulation while performing the Sternberg WM task under threat of shock (Substudy 2).

Study population: The study population will consist of up to 184 healthy volunteers between the ages of 18-50.

Design: This study will consists of two (sub-studies 1 and 2) or three (sub-study 3) outpatient visits (1 MRI, 1 or 2 TMS visits [2 for sub-study 3]). In this protocol we will explore the effect of TMS in three sub-studies in the TMS study visit. The sub-studies will contain either the NPU or the Sternberg task during the TMS visits. The first visit (MRI) will consist of the same procedures for all sub-studies. Each subject will be assigned to only one of the sub-studies.

Sternberg Task: Expose subjects to active or sham TMS to a region of the frontoparietal attention network during the Sternberg WM task. Subjects will have to maintain a series of letters in WM for a brief interval during blocks of safety and threat of shock.

NPU Task: Expose subjects to active or sham TMS to a region of the frontoparietal attention network during the NPU threat test. Subjects will be exposed to blocks in which they are either 1) safe from shock (neutral), 2) at risk of shock delivered only during a cue (predictable), or 3) at risk of shock presented randomly (unpredictable).

Outcome measures: In both studies the primary outcome measure will be anxiety-potentiated startle (APS), which is the increase in startle magnitude during periods of threat compared to periods of safety. We expect active, but not sham TMS to increase activity in the dlPFC, and therefore reduce APS in both studies

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ages 18-50
* Subjects able to give their consent
* Right handed

EXCLUSION CRITERIA:

* Non-English speaking individual
* Any significant medical or neurological problems (e.g. cardiovascular illness, respiratory illness, neurological illness, seizure, etc.)
* Current or past Axis I psychiatric disorder(s) as identified with the Structured Clinical Interview for DSM-IV, non-patient edition (SCID-np)
* Active or history of active suicidal ideation.
* Evidence of a first-degree relative with history of psychosis or bipolar disorder; specifically, participant will know diagnosis or treatment in order to confirm presence of disorder.
* Alcohol/drug problems in the past year or lifetime alcohol or drug dependence according to the Structured Clinical Interview for DSM-IV.
* Current use of medications that act on histamine (i.e. diphenhydramine), dopamine (methylphenidate), norepinephrine (buproprion), serotonin (sertraline), or acetylcholine (amitryptiline) receptors. Subjects will be excluded on this basis if they either 1) take these medications on a chronic basis, or 2) if they have taken the drug within 5 half-lives of the drug metabolism, determined by the medical professional at the time of screening.
* History of seizure (childhood febrile seizures are acceptable and these subjects may be included in the study),
* History of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold (table below).
* Pregnancy, or positive pregnancy test.
* Neurological syndrome of the arm (e.g., carpal tunnel syndrome, cubital tunnel syndrome, etc.)
* Positive urine toxicology screen during the screening visit.
* IQ <80
* Employee or staff of NIMH or are an immediate family member of a NIMH employee, staff, or NIMH contractors.
* Allergy to lidocaine or topical anesthetics (participants in sub-study 3 only).
* Any medical condition that increases risk for fMRI or TMS:

  * Any metal in their body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if you were a welder or metal worker, since you may small metal fragments in the eye.
  * Participants who are uncomfortable in small closed spaces (have claustrophobia) and would feel uncomfortable in the MRI machine
  * Patients who have difficulty lying flat on their back for up to 60 min in the scanner
  * History of hearing loss

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grillon, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Balderston NL, Quispe-Escudero D, Hale E, Davis A, O'Connell K, Ernst M, Grillon C. Working memory maintenance is sufficient to reduce state anxiety. Psychophysiology. 2016 Nov;53(11):1660-1668. doi: 10.1111/psyp.12726. Epub 2016 Jul 19. PMID 27434207
- [Background] Schmitz A, Grillon C. Assessing fear and anxiety in humans using the threat of predictable and unpredictable aversive events (the NPU-threat test). Nat Protoc. 2012 Feb 23;7(3):527-32. doi: 10.1038/nprot.2012.001. PMID 22362158
- [Background] Slotema CW, Blom JD, Hoek HW, Sommer IE. Should we expand the toolbox of psychiatric treatment methods to include Repetitive Transcranial Magnetic Stimulation (rTMS)? A meta-analysis of the efficacy of rTMS in psychiatric disorders. J Clin Psychiatry. 2010 Jul;71(7):873-84. doi: 10.4088/JCP.08m04872gre. Epub 2010 Mar 9. PMID 20361902
- [Derived] Balderston NL, Roberts C, Beydler EM, Deng ZD, Radman T, Luber B, Lisanby SH, Ernst M, Grillon C. A generalized workflow for conducting electric field-optimized, fMRI-guided, transcranial magnetic stimulation. Nat Protoc. 2020 Nov;15(11):3595-3614. doi: 10.1038/s41596-020-0387-4. Epub 2020 Sep 30. PMID 33005039
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-M-0042.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Substudy 1 Active and Sham; Substudy 2 Active and Sham: HVs that receive active and sham TMS over the right dlPFC
  Transcranial Magnetic Stimulation Sham: TMS device is used to determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects.
  Transcranial Magnetic Stimulation: TMS device is used to determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects.
Period: Overall Study
Arm/Group | Substudy 1 Active and Sham | Substudy 2 Active and Sham | Substudy 3 Active and Sham
Started | 28 | 0 | 26
Completed | 19 | 0 | 20
Not Completed | 9 | 0 | 6

BASELINE CHARACTERISTICS:
Population: No participants were recruited in Substudy 2. Study was stopped because lead investigator (Dr. Balderston) changed position prior to the initiation of Study 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Substudy 1 Active and Sham | Substudy 2 Active and Sham | Substudy 3 Active and Sham | Total
Number analyzed (Participants) | 28 | 0 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 28 |  | 26 | 54
  >=65 years | 0 |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.25 (7.414392375) |  | 30.46153846 (8.52701936) | 28.7962963 (8.129460894)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 |  | 16 | 31
  Male | 13 |  | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 |  | 3 | 7
  Not Hispanic or Latino | 24 |  | 23 | 47
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 5 |  | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 4 |  | 5 | 9
  White | 16 |  | 12 | 28
  More than one race | 3 |  | 1 | 4
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 |  | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Anxiety-potentiated Startle
Description: Electromyography Facial electromyography (EMG) startle responses were recorded from the left orbicularis oculi muscle at 2000 Hz using a Biopac MP160 unit (Biopac; Goleta, CA) via 15 × 20 mm hydrogel coated vinyl electrodes (Rhythmlink #DECUS10026; Columbia, SC).
  Startle EMG was bandpass filtered from 30 to 300 Hz, rectified, and smoothed using a 20-ms sliding window. Startle responses were scored as the peak (max during the 20 ms to 120 ms post-noise window) - the baseline (50 ms pre-noise window), and converted to t-scores with a mean of 50 and a standard deviation of 10 (tx = [Zx × 10] + 50). Greater t-scores mean larger blinks, which could be associated with greater anxiety, however there is no clinically relevent threshold. Noisy trials (baseline SD > 2x run SD) were excluded, and "no blink" (peak < baseline range) trials were coded as 0. To calculate APS, we subtracted the response during the neutral ITI from the response during the unpredictable ITI.
Time Frame: Pre and post stimulation
Population: Healthy Volunteers
Measure: Mean (Standard Error); unit: T-scores
Arm/Group | Substudy 1 Active and Sham | Substudy 3 Active and Sham
Number analyzed (Participants) | 19 | 19
T-scores
  Active | 6.032164105 (1.31706568) | 2.420193836 (1.174992336)
  Sham | 3.412441384 (1.02011584) | 4.467812115 (0.966471881)
  No TMS / Pre-stimulation | 2.832028871 (0.989278736) | 4.960918182 (1.111076546)

2. Primary Outcome: Working Memory (WM) Related Anxiety Downregulation While Performing the Sternberg WM Task Under Threat of Shock.
Description: Sternberg Task: Expose subjects to active or sham TMS to a region of the frontoparietal attention network during the Sternberg WM task. Subjects will have to maintain a series of letters in WM for a brief interval during blocks of safety and threat of shock.
  Electromyography Facial electromyography (EMG) startle responses are recorded from the left orbicularis oculi muscle at 2000 Hz.
  Startle EMG is bandpass filtered from 30 to 300 Hz, rectified, and smoothed using a 20-ms sliding window. Startle responses are scored as the peak (max during the 20 ms to 120 ms post-noise window) - the baseline (50 ms pre-noise window), and converted to t-scores (tx = [Zx × 10] + 50). Noisy trials (baseline SD > 2x run SD) are excluded, and "no blink" (peak < baseline range) trials are coded as 0. These t scores are then averaged across trials within each condition, and threat-safe contrasts are calculated independently for each level of load (low vs. high) and timing (maintenance vs. ITI).
Time Frame: Pre and post stimulation
Population: as for baseline characteristics
Groups:
- Substudy 2: HVs that receive TMS over the right dlFPC
  Transcranial Magnetic Stimulation Sham: TMS device is used to determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects.
  Transcranial Magnetic Stimulation: TMS device is used to determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects.
Arm/Group | Substudy 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: During study participation, which typically lasted less than 1 month.
Description: The Principal Investigator was responsible for detecting, documenting, and reporting unanticipated problems, adverse events (AEs), including serious adverse events (SAEs), and deviations in accordance with NIH policy, IRB requirements, and federal regulations. Relatedness to the research of all serious adverse events will be determined by the PI in consultation with the CD.
Groups:
- Substudy 3: HVs will receive offline TMS to the lest IPS (FPN)
  Transcranial Magnetic Stimulation: TMS device is used to determine the effect of non-invasive brain stimulation on anxiety and anxiety-cognition interactions in healthy subjects.
Arm/Group | Substudy 1 Active and Sham | Substudy 2 Active and Sham | Substudy 3
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/0 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/0 | 0/26
Other Adverse Events (participants affected / at risk) | 8/28 | 0/0 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1 Active and Sham (N=28) | Substudy 2 Active and Sham (N=0) | Substudy 3 (N=26)
Possible vasovagal syncope (Product Issues) | 1 (1) | 0 (0) | 0 (0) — Unexpected adverse event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1 Active and Sham (N=28) | Substudy 2 Active and Sham (N=0) | Substudy 3 (N=26)
mild headache (Product Issues) | 4 (5) | 0 (0) | 3 (3)
scalp or face discomfort (Product Issues) | 3 (3) | 0 (0) | 0 (0)
non-medical device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) — computer malfunction resulting in mild unexpected shock presentation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT03027414/Prot_SAP_002.pdf
  • Informed Consent Form (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT03027414/ICF_001.pdf